CLINICAL TRIAL: NCT00595075
Title: Effects of Ramelteon on Sleep and Neurobehavioral Performance in a Simulated Night Shift Preceded by a Sleep Opportunity
Brief Title: Ramelteon for a Nap Prior to a Night Shift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Elizabeth B. Klerman, Associate Professor, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Takeda - 103113
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: sleep; performance; night shift; Ramelteon; Healthy Individuals
MeSH Terms: interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ramelteon 8 mg will be given once prior to a 2-hour nap
  Interventions: Drug: Ramelteon
- 2 (Placebo Comparator): Placebo will be given once prior to a 2-hour nap
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8 mg tablet by mouth x 1 dose
  Other Names: Rozerem
  Arms: 1
Drug: placebo — placebo identical in appearance to active experimental drug x 1 dose
  Arms: 2

SUMMARY:
Night shift-workers are often advised to take a prophylactic nap prior to starting the shift in order to improve alertness and performance. However, individuals often report difficulty initiating and maintaining sleep at that time of the day secondary to the alerting influence of the near-24 hour circadian rhythm (biological clock). A sleep-promoting medication may improve the quality of an evening nap and subsequent alertness and performance during a night shift. We will use Ramelteon, a melatonin agonist that is FDA approved for insomnia, in order to test the following hypotheses:

1. ramelteon, compared with placebo, will significantly increase sleep efficiency during a 2-hour nap;
2. sleep inertia, as assessed by neurobehavioral tests and subjective and objective sleepiness assessments will not be significantly increased after ramelteon treatment compared with placebo treatment; and
3. neurobehavioral performance, subjective and objective sleepiness, and subjective mood during a simulated 8-hour night shift will be significantly improved when ramelteon is given prior to a prophylactic nap compared to a prophylactic nap with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years;
* Non-smoking for at least 6 months;
* Healthy (no medical, psychiatric or sleep disorders);
* No clinically significant deviations from normal in medical history, vital signs, physical examination, blood chemistry and hematology, and ECG;
* Women of childbearing potential must agree to use an acceptable method of birth control, and must have a negative serum pregnancy test;
* Body mass index of > 18 or < 30 kg/m∧2;
* No drugs or medication likely to affect sleep or alertness, as determined by the investigators;
* Habitual caffeine consumption < 300 mg per day on average;
* Habitual alcohol consumption < 10 alcoholic units per week on average.

Exclusion Criteria:

* History of alcohol or substance abuse;
* Positive result on drugs of abuse screening;
* Current or past history of sleep disorders, including but not limited to obstructive sleep apnea, or any significant sleep complaint;
* Psychiatric disorder, including a history of depression or dysthymia (characterized by depressed mood on the majority of days for at least two years);
* Recent acute or chronic medical disorder, including but not limited to hepatic impairment and severe chronic obstructive pulmonary disease;
* History of intolerance or hypersensitivity to melatonin or melatonin agonists;
* Pregnancy or lactation;
* Shift work;
* Transmeridian travel (2 or more time zones) in past 2 months;
* Any other scientific or medical reason, as determined by the PI, such as non-compliance with protocol or intolerance to inpatient study conditions.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2007-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shantha Rajaratnam, PhD, Principal Investigator — Brigham and Women's Hosptial; Elizabeth B Klerman, MD,PhD, Principal Investigator — Brigham and Women's Hospital

REFERENCES:
- [Result] Cohen DA, Wang W, Klerman EB, Rajaratnam SM. Ramelteon prior to a short evening nap impairs neurobehavioral performance for up to 12 hours after awakening. J Clin Sleep Med. 2010 Dec 15;6(6):565-71. PMID 21206545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited
Pre-assignment Details: Participants received 1 dose of ramelteon or placebo during the first inpatient visit and then returned approximately four weeks later for the other condition, counterbalanced for order
Groups:
- Ramelteon in First Crossover Period: Ramelteon 8 mg will be given prior to a 2-hour nap
- Placebo in First Crossover Period: Placebo will be given prior to a 2-hour nap
Period: Overall Study
Arm/Group | Ramelteon in First Crossover Period | Placebo in First Crossover Period
Started | 6 | 5
Completed | 5 | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon in First Crossover Period | Placebo in First Crossover Period | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22.7 (4.1) | 26.8 (3.2) | 24.5 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency
Description: total sleep time/time in bed * 100% (higher values indicate better outcome)
Time Frame: 2 hours
Population: All participants that completed both crossover periods
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Ramelteon: Ramelteon 8 mg will be given prior to a 2-hour nap
- Placebo: Placebo will be given prior to a 2-hour nap
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 10 | 10
percent | 89.1 (9.8) | 83.3 (14.3)

2. Other Pre Specified Outcome: Post-nap Assessment - Visual Analog Scale
Description: numerical scale of increasing alertness from 0-100 (higher values are better outcome)
Time Frame: 71 minutes
Population: All participants that completed both crossover periods
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | 61.1 (18.6) | 67.1 (22.8)

3. Other Pre Specified Outcome: Post Nap Assessment - Karolinska Sleepiness Scale
Description: numerical scale of increasing sleepiness from 1-9 (higher values indicate worse outcome)
Time Frame: 71 minutes
Population: All participants that completed both crossover periods
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | 5.4 (1.6) | 4.8 (1.8)

4. Other Pre Specified Outcome: Post Nap Assessment - Digit Symbol Substitution Test (Correct Answers)
Description: A cognitive throughput task consisting of matching symbols to numerical keys; higher numbers indicate a better score
Time Frame: 71 minutes
Population: All participants that completed both crossover periods
Measure: Mean (Standard Deviation); unit: correct answers
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 10 | 10
correct answers | 50.4 (9.3) | 53.3 (9.3)

5. Other Pre Specified Outcome: Post Nap Assessment - Karolinska Drowsiness Test
Description: EEG spectral analysis of 5.5-9.0 Hz frequency activity (theta low-frequency alpha), with higher activity indicating increased drowsiness and worse outcome
Time Frame: 71 minutes
Population: All participants completing both crossover periods
Measure: Mean (Standard Deviation); unit: microvolts^2/Hz
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 10 | 10
microvolts^2/Hz | 4.9 (4.5) | 4.0 (5.6)

6. Other Pre Specified Outcome: Psychomotor Vigilance Task - Median Reaction Time
Description: Visual-motor reaction time in which participants hit a button on a response box as fast as possible in response to a visual target (lower values indicate better outcome)
Time Frame: 8 hours
Population: All participants completing both crossover periods
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 10 | 10
seconds | 0.662 (0.16) | 0.362 (0.25)

7. Other Pre Specified Outcome: Psychomotor Vigilance Task - Number of Lapses
Description: Number of trials per test battery with a reaction time >0.5 seconds (higher values indicate worse outcome)
Time Frame: 8 hours
Population: All participants completing both crossover periods
Measure: Mean (Standard Deviation); unit: lapses
Arm/Group | Ramelteon | Placebo
Number analyzed (Participants) | 10 | 10
lapses | 15.5 (16.3) | 13.2 (16.0)

ADVERSE EVENTS:
Time Frame: During each 28-hr inpatient study admission
Arm/Group | Ramelteon | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
Circadian phase was not measured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less